CLINICAL TRIAL: NCT03885687
Title: Exercise With Music Program for ICU Survivors
Brief Title: Exercise With Music for ICU Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Zhan Liang, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180508
Record Dates: First submitted 2018-12-06; First posted 2019-03-22 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Critical Illness; Intensive Care Unit Syndrome
Keywords: Rehabilitation; Exercise; Music Intervention
MeSH Terms: conditions — Critical Illness; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise with Music Intervention (Experimental): The Exercise with Music intervention is a recorded exercise playlist, which is tailored to a patient's individual physical abilities and music choices.
  Interventions: Behavioral: Exercise with Music
- Active Control Group (Active Comparator): The active control group will receive exercise brochure and will be advised to exercise at least twice daily.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise with Music — The Exercise with Music intervention is recorded exercise playlist, which provide exercise instructions tailored to patients' musical choices and exercise capacity.
  Arms: Exercise with Music Intervention
Behavioral: Exercise — The exercise group will receive exercise brochure and will be advised to exercise at least twice daily.
  Arms: Active Control Group

SUMMARY:
This project will test whether the individualized music-enhanced exercise playlist (Exercise with Music intervention) can prevent further physical and psychological deterioration and motivate ICU survivors to more actively participate in their rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* length of ICU stay >5 days (excludes patients with less comorbidity)
* within 72 hours of ICU discharge (standardizes time to begin intervention)
* ability to independently move upper and lower extremities (required to participate in intervention)
* ability to speak English or Spanish

Exclusion Criteria:

* documented mental incompetence
* dependent status pre-ICU admission (KATZ, activity daily living scale)
* evidence of delirium using the Confusion Assessment Method (CAM)
* hearing impairment
* documented "comfort measures only" in the electronic medical record
* prior residence in a long-term care facility
* unstable hemodynamics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | One year
  Number of subjects enrolled into the study divided by number of subjects approached X 100%
Acceptability of intervention as measured by a questionnaire | Day five
  A self-designed 8-item questionnaire is administered to assess subjects' feedback regarding the intervention. Five questions are likert-scale questions (strongly disagree, disagree, undecided, agree, strongly agree); three questions are yes or no questions. If the results of the questionnaire show that majority of patients answer "agree or strongly agree" and "yes", this would indicate that the intervention is acceptable. If the results of the questionnaire show that majority of the patients answer "strongly disagree or disagree" and "no", this would indicate that the intervention is not acceptable.
Number of participants that complete the intervention as prescribed | Day 5
  Count of participants who exercise twice daily for five days (upper and lower extremity exercise). Each session includes five movements. The number of movements and sessions of the intervention delivered within and beyond the 5-day mandatory regimen will be documented.
Number of participants that complete the intervention beyond the 5-day mandatory sessions | Day 11
  Count of participants who complete additional exercise sessions beyond the prescribed exercise regimen (twice daily for five days). Each session includes five movements.
Number of participants with adverse events | Day 5
  Adverse events are any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the trial intervention.

SECONDARY OUTCOMES:
Effect size of the Exercise with Music intervention | One year
  Estimated effect size of the intervention on outcome measures to calculate sample size for a larger future study.
Changes in activity | Baseline, Day 5
  Activity will be monitored using an Actiwatch (Philips Respironics) placed on subjects' wrists at enrollment. The Actiwatch is a small, lightweight, limb-worn activity monitoring device. It contains an accelerometer that is capable of sensing any motion with minimal acceleration of 0.01g to measure long-term gross motor activity and intensity of motion.
Changes grip strength | Baseline, Day 5
  Grip strength will be assessed using handgrip dynamometer.
Changes grip strength at hospital discharge | Day 5, Day 11
  Grip strength will be assessed using handgrip dynamometer.
Changes in Foot Strength | Baseline, Day 5
  Foot strength will be assessed objectively using hand-held dynamometer.
Changes in Foot Strength at hospital discharge | Day 5, Day 11
  Foot strength will be assessed objectively using hand-held dynamometer.
Changes in Motivation (Visual Analog Scale) | Baseline, Day 5
  Motivation will be measured by the visual analog scale (VAS) with scores from 0 to 100. "0" indicates "not motivated to do exercise at all"; "100" indicates "extremely motivated to do exercise".
Changes in Motivation (Visual Analog Scale) at hospital discharge | Day 5, Day 11
  Motivation will be measured by the visual analog scale (VAS) with scores from 0 to 100. "0" indicates "not motivated to do exercise at all"; "100" indicates "extremely motivated to do exercise".
Changes in Anxiety (Visual Analog Scale) | Baseline, Day 5
  Anxiety will be measured by the visual analog scale (VAS) with scores from 0 to 100. "0" indicates "no anxiety"; "100" indicates "extremely anxious".
Changes in Anxiety (Visual Analog Scale) at hospital discharge | Day 5, Day 11
  Anxiety will be measured by the visual analog scale (VAS) with scores from 0 to 100. "0" indicates "no anxiety"; "100" indicates "extremely anxious".
Changes in Anxiety (NIH Toolbox) | Baseline, day 5
  Anxiety will also be assessed using the NIH Toolbox Emotion Battery (fear-affect survey), CAT format. Each item administered has a 5-point scale with options ranging from "never" to "always." The survey is scored using IRT methods. Higher scores are indicative of more feelings of anxiety.
Changes in Anxiety (NIH Toolbox) at hospital discharge | Day 5, Day 11
  Anxiety will also be assessed using the NIH Toolbox Emotion Battery (fear-affect survey), CAT format. Each item administered has a 5-point scale with options ranging from "never" to "always." The survey is scored using IRT methods. Higher scores are indicative of more feelings of anxiety.
Changes in Depression (NIH Toolbox) | Baseline, Day 5
  Depression will be assessed using the NIH Toolbox Emotion Battery (sadness survey), CAT format. Each item administered has a 5-point scale with options ranging from "never" to "always" (adults) or "almost always". higher scores are indicative of more depressive.
Changes in Depression (NIH Toolbox) at hospital discharge | Day 5, Day 11
  Depression will be assessed using the NIH Toolbox Emotion Battery (sadness survey), CAT format. Each item administered has a 5-point scale with options ranging from "never" to "always" (adults) or "almost always". higher scores are indicative of more depressive.

CONTACTS AND LOCATIONS:
Overall Officials: Zhan Liang, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang Z, Munro C, Yip H, Ji M, Sena Moore K, Ferreira T, Signorile JF, Pan Y. Randomized Controlled Study of Self-Managed Music-Guided Exercise Intervention Following Intensive Care. Nurs Res. 2023 May-Jun 01;72(3):193-199. doi: 10.1097/NNR.0000000000000644. Epub 2023 Jan 9. PMID 36638206
- [Derived] Liang Z, Yip H, Sena Moore K, Ferreira T, Ji M, Signorile JF, Munro C. Self-Managed Music-Guided Exercise Intervention Improved Upper and Lower Extremity Muscle Strength for ICU Survivors-A Pilot Randomized Controlled Study. Biol Res Nurs. 2022 Apr;24(2):145-151. doi: 10.1177/10998004211050297. Epub 2021 Nov 5. PMID 34738474